CLINICAL TRIAL: NCT04122404
Title: Point-of-care Strategies to Improve Tuberculosis Care Among Severely Immunosuppressed HIV-infected Patients
Brief Title: POC Strategies to Improve TB Care in Advanced HIV Disease
Acronym: TBPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); National Tuberculosis Control Programme, Ghana (Unknown); Odense Patient Data Explorative Network (Other); University of Ghana (Other); Tema General Hospital, Ghana (Unknown); Lekma Hospital, Ghana (Unknown); Korle-Bu Teaching Hospital, Ghana (Unknown)
Responsible Party: Principal Investigator, Johanna Maria Åhsberg, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: OP_861
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Extrapulmonary Tuberculosis; Tuberculosis, Pulmonary; Human Immunodeficiency Virus (HIV); Acquired Immunodeficiency Syndrome
Keywords: Point-of-care systems; Tuberculosis/Diagnosis; Biomarkers/Urin; Lipopolysaccharides/urine; Audit intervention; Diagnostic tests/Routine; Ultrasound; Bedside; Biobank; Stepped wedge cluster randomised trial; Multicenter study; Audit and feedback; Ghana; Adult; Hospitalization
MeSH Terms: conditions — Tuberculosis, Extrapulmonary; Tuberculosis, Pulmonary; Acquired Immunodeficiency Syndrome; Tuberculosis; Disease

STUDY DESIGN:
Intervention Model Description: Open label multi-center stepped wedge cluster-randomized controlled implementation trial of the use of urine-based LF-LAM in addition to routine sputum-based TB diagnostic tests to guide initiation of TB treatment among adult hospitalized patients with advanced HIV. The design offers a randomised method of evaluation of the intervention at cluster level. Applying the stepped wedge design ensures that all participating HIV/ART clinic attached wards will have received the intervention at the end of the study period, and provides the basis for the LF-LAM test to become an integrated part of TB health care services also after the project finishes. Clinic staff will be trained on how to use and interpret the LF-LAM test and in TB diagnostic guidelines as outlined by WHO. An Audit and feedback study will identify leaky steps in the TB diagnostic pathway and further strengthen the implementation and possible impact of the LF-LAM test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Routine TB diagnostic care (sputum smear microscopy, sputum Xpert MTB/Rif / sputum Xpert MTB/Rif Ultra, sputum culture) + Intervention
  Intervention: LF-LAM is made available at the study site for the clinical staff to use; Training of clinical staff in national TB guidelines and LF-LAM use together with staff from the National TB Programme in Ghana
  Interventions: Diagnostic Test: LF-LAM
- Standard of care (No Intervention): Routine TB diagnostic care (sputum smear microscopy, sputum Xpert MTB/Rif / sputum Xpert MTB/Rif Ultra, sputum culture)

INTERVENTIONS:
Diagnostic Test: LF-LAM — Open label multi-center stepped wedge cluster-randomized controlled trial with implementation of LF-LAM. All clusters (i.e. HIV/ART clinic attached wards) start with standard of care and are then randomized to switch to the intervention phase at predefined time points.
  Other Names: Lateral flow urine lipoarabinomannan assay; Determine TM TB LAM Ag test
  Arms: Intervention

SUMMARY:
Tuberculosis (TB) remains the major cause of morbidity and mortality among patients with HIV. Sub-optimal diagnostics contributes towards poor patient outcome and there is an urgent need to identify non-sputum-based point-of-care diagnostic tests. The urine based lateral flow lipoarabinomannan TB diagnostic test (LF-LAM) is a simple, inexpensive point-of-care test. In 2015, the World Health Organization endorsed LF-LAM for conditional use among patients with advanced HIV, but uptake of the test in clinical practices has been poor.

The investigators aim to identify point-of-care (POC) strategies that can improve TB case detection and clinical outcomes among patients with advanced HIV. The project includes a main study and two sub-studies.

The main study is a multicenter stepped wedge cluster-randomized controlled trial of LF-LAM implementation among patients with advanced HIV with 8-weeks follow-up. LF-LAM will be added to standard care and implemented stepwise at three hospitals in Ghana. Education in national TB treatment guidelines in collaboration with the Tuberculosis Control programme in Ghana, and Clinical audit of clinical staff with feedback, will be used to assess and strengthen LF-LAM implementation. The primary outcome time to TB treatment, for which a sample size of 690 participants will provide >90% power to detect a minimum of 7 days reduction. Secondary outcomes are: TB related morbidity, TB case detection, time to TB diagnosis and overall early mortality at 8 weeks. The HIV-associated TB epidemiology including genotypic analyses of M. tuberculosis isolates obtained through the main study will be described. In sub study A, focused ultrasound of lungs, heart and abdomen will be performed in a sub cohort of 100 participants. In sub study B, the investigators will establish a biobank and data warehouse for storage of blood, urine and sputum samples collected from participants that enter the study at Korle-Bu Teaching hospital.

It is expected that LF-LAM will lead to earlier diagnosis and treatment of TB. Findings may further guide scaling-up of LF-LAM. The HIV-associated epidemic including genotypic properties and resistance properties which is important for improved management will be detailed. The investigators further expect to evaluate the potential of bedside ultrasound as a clinical tool in management of HIV/TB co-infected patients. The unique Ghanaian HIV-cohort and biobank may facilitate rapid evaluation of future prognostic biomarkers and new point-of-care TB diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* 18 years and above
* Able to give informed consent
* Admitted at the wards attached to the research site ART/HIV-clinic
* Eligible for LF-LAM testing (defined by WHO in the LF-LAM policy update 2019): CD4-cell-count ≤200 cells/μL (the last measured CD4-cell-count); or a WHO clinical stage 3 or 4 event at presentation for care; or seriously ill defined by WHO (respiratory rate > 30/min, temperature > 39°C, heart rate > 120/min or unable to walk unaided); or a positive WHO TB symptom screening including one of the following symptoms: current cough, fever, weight loss, or night sweats

Exclusion Criteria:

* Anti-tuberculous treatment including preventive treatment with Isoniazide within the last 60 days
* Earlier participation in the same study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Time to TB treatment initiation | 8 weeks follow up
  Time to TB treatment initiation defined by time from TB diagnosis suspected to start of anti-tuberculous treatment provided.

SECONDARY OUTCOMES:
TB related morbidity | 8 weeks follow up
  The difference in the proportion of TB patients with reduced TB morbidity score at 8 weeks follow up using "The Bandim tuberculosis score" with grading 0-13, where a reduction in the score may be used as a measurement of clinical improvement.
TB case detection | 8 weeks follow up
  Defined as proportion of patients with (i) microbiologically confirmed TB diagnosis and (ii) clinically confirmed TB diagnosis
Time to TB diagnosis | 8 weeks follow up
Time to all-cause mortality. | 8 weeks follow up
  Mortality rates during follow up. Underpowered

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Åhsberg, MD, Principal Investigator — Dept. of Infectious Diseases, Odense University Hosp., Univ. of Southern Denmark; Isik Somuncu Johansen, Prof, Study Director — Dept. of Infectious Diseases, Odense University Hosp., Univ. of Southern Denmark; Margaret Lartey, Prof, Study Chair — School of Medicine and Dentistry, University of Ghana; Stephanie Bjerrum, MD, Study Chair — Dept. of Infectious Diseases, Odense University Hosp., Univ. of Southern Denmark; Åse Bengaard Andersen, Prof, Study Chair — Dept. of Infectious Diseases, Odense University Hosp., Univ. of Southern Denmark; Ernest Kenu, MD, Study Chair — Dept. of Epidemiology and Disease Control, Univ. of Ghana
Locations (3):
- Ghana (3):
  - Korle Bu Teaching Hospital, Accra
  - Tema General Hospital, Tema
  - Lekma Hospital, Teshie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229